CLINICAL TRIAL: NCT01648478
Title: Evaluation of Plasma IRAP Secreted Protein as a New Insulin Sensitivity Biomarker, Using Hyperinsulinemic Euglycemic Clamp
Brief Title: IRAPs (Secreted Insulin Regulated AminoPeptidase): a New Insulin Sensitivity Biomarker
Acronym: IRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Cisbio Bioassays (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011.705
Record Dates: First submitted 2012-06-27; First posted 2012-07-24 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Insulin Resistance
Keywords: IRAP; insulin sensitivity marker
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Other: It is a hyperinsulinemic-euglycemic clamp.

INTERVENTIONS:
Other: It is a hyperinsulinemic-euglycemic clamp. — The hyperinsulinemic-euglycemic clamp includes three periods:
  * A basal period (from T-30 to T0)
  * The infusion of insulin at a constant rate (first level at 1 mUI.kg-1.min-1 and a second level at 2 mUI.kg-1.min-1) during 4 hours ( to obtain stable hyperinsulinemia)
  * The infusion of glucose at variable rate (so as to maintain euglycemia)

SUMMARY:
Previous studies have demonstrated defects in the trafficking and translocation of GLUT4 glucose transporter in skeletal muscle and adipose tissue to be a major cause of insulin resistance in humans. IRAP (Secreted Insulin Regulated AminoPeptidase) is a protein which collocalizes and is translocated with GLUT4 to the plasma membrane in response to insulin. The extracellular domain of IRAP is cleaved and released in the bloodstream.

Therefore, IRAP plasma concentration could be a good marker of insulin sensitivity.

In this study the investigators seek to confirm this hypothesis by using the gold standard of insulin sensitivity assessment: the hyperinsulinemic-euglycemic clamp.

It is a multicenter descriptive study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (sex ratio = 1)
* Aged from 18 to 35 years
* Fasting glycemia < 6mmol/L
* Total cholesterol < 7mmol/L
* Triglycerides < 1.5 mmol/L
* CRPus < 5 mg/L
* Creatinine clearance < 80mL/min according to Cockroft formula
* Liver enzymes (ALanine AminoTransférase and ASpartate AminoTransférase) < 1.5 times normal values

Exclusion Criteria:

* Subject not in compliance with the recommendations of French National Law in force
* Medical history of metabolic disease (diabetes, dyslipidemia), endocrine disease, renal insufficiency
* Drug use that could affect glucose metabolism and the renin angiotensin aldosterone system
* Blood pressure > 140/90mmHg
* Tea and coffee consumption more than 5 cups per day
* Subject who smoke more than 5 cigarettes per day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
IRAP plasma concentration during the hyperinsulinemic euglycemic clamp | 30 min before the clamp and during the clamp every 10 min for a duration of 240 min.
  Enzyme-linked Immunosorbsent assay (Sandwich ELISA)

SECONDARY OUTCOMES:
Glucose Infusion Rate (GIR) | at T90, T100, T110, T120 minutes and T210, T220, T230, T 240 minutes
  It is an average rate of glucose infused at steady state of the first and second level of insulinemia infusion
Oxydative stress markers | at T0, T120 and T240 min
  TBARS, GSH, GSSG and nitroalbumin assessments

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, Pr, Principal Investigator — Centre de recherche en nutrition humaine Rhone-Alpes
Locations (1):
- Centre de recherche en nutrition humaine Rhone-Alpes, Pierre-Bénite, France

REFERENCES:
- [Background] Trocme C, Gonnet N, Di Tommaso M, Samouda H, Cracowski JL, Cracowski C, Lambert-Porcheron S, Laville M, Nobecourt E, Gaddhab C, Le Lay A, Bohn T, Poitou C, Clement K, Al-Mulla F, Bitar MS, Bottari SP. Serum IRAP, a Novel Direct Biomarker of Prediabetes and Type 2 Diabetes? Front Mol Biosci. 2021 Feb 16;7:596141. doi: 10.3389/fmolb.2020.596141. eCollection 2020. PMID 33665204
- See also: Related Info — http://www.crnh-rhone-alpes.fr